CLINICAL TRIAL: NCT01543737
Title: Single-blind Randomised Pragmatic Trial Comparing the Effectiveness of Two Hyaluronic Acid Viscosupplements, DUROLANE® (Single Injection) Versus HYALGAN® (Three Injections) for Symptomatic Tibiofemoral Osteoarthritis of the Knee.
Brief Title: Effectiveness of Two Hyaluronic Acids in Osteoarthritis of the Knee
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: post transfer of company ownership from Smith & Nephew to Bioventus LLC
Sponsor: Bioventus LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SNOF EC 01/2010
Record Dates: First submitted 2012-02-20; First posted 2012-03-05 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single injection hyaluronic acid (Active Comparator): 3ml hyaluronic acid (DUROLANE)
  Interventions: Device: 3ml hyaluronic acid (DUROLANE)
- Three injection hyaluronic acid (Active Comparator): 2ml hyaluronic acid (HYALGAN)
  Interventions: Device: 2ml hyaluronic acid, (HYALGAN)

INTERVENTIONS:
Device: 3ml hyaluronic acid (DUROLANE) — DUROLANE Hyaluronic acid 20mg/ml
  Arms: Single injection hyaluronic acid
Device: 2ml hyaluronic acid, (HYALGAN) — HYALGAN Hyaluronic acid 10mg/ml
  Arms: Three injection hyaluronic acid

SUMMARY:
The purpose of this study is to assess whether a single injection hyaluronic acid (HA) product is not inferior to a 3 injection HA product at 24 weeks (6 months), in terms of effectiveness in reducing pain when walking in patients suffering from symptomatic tibiofemoral osteoarthritis of the knee.

DETAILED DESCRIPTION:
non-inferiority study of two HA products commercially availalble

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 and < 85
* Tibiofemoral osteoarthritis of the knee according to the American College of Rheumatology clinical criteria, in the Kellgren-Lawrence (KL) stages II-III, confirmed by radiology (< 3 months)
* Unilateral symptomatic osteoarthritis of the knee causing pain when walking (WOMAC A1 scale), assessed over the previous 24 hours on a scale of 0 to 10: Pain when walking: ≤ 3 and < 8
* Bilateral osteoarthritis of the knee, if pain in the other knee is < 3 (10-point numerical scale)
* Patient: outpatient, capable of walking 50 metres without a walking stick, crutches or a walker, capable of reading, understanding, signing and dating the patient information sheet
* Patient with social security cover

Exclusion Criteria:

* Osteoarthritis of the knee in Kellgren-Lawrence (KL) stages I and IV
* Bilateral symptomatic osteoarthritis of the knee causing pain when walking (WOMAC A1 scale), assessed on a scale of 0 to 10: Pain when walking > 3, in both knees
* Predominant symptomatic patellofemoral osteoarthritis of the knee
* Congestive manifestation of osteoarthritis of the knee defined according to the Knee Osteoarthritis Flare-Ups Score (KOFUS) criteria
* Last viscosupplementation of the affected knee < 6 months before, last injection of corticosteroids < 2 months before
* Known hypersensitivity to avian proteins and hyaluronic acids;
* History of joint replacement or major surgery in the affected knee in the last six months
* History of arthroscopy or surgery in the affected knee in the last three months
* Symptomatic hip disease on the same side or other side of the body
* Joint replacement or any other surgery planned in the next six months
* History of septic arthritis of the affected knee
* Skin complaint affecting the knee at the injection site
* Haemorrhagic disease contraindicating, in the doctor's opinion, any intra-articular injection
* In order to respect the pragmatic nature of the study:
* Any medical and / or pathological condition that, in the investigator's opinion, makes the subject unsuitable for inclusion
* Any medical and / or pathological condition that, in the investigator's opinion, would be a contraindication for an intra-articular injection
* Any other complaint that, in the investigator's opinion, would impede the assessment of the effectiveness of the affected knee
* Any treatment administered to the patient that may interfere with the interpretation of the study results
* Use of glucocorticosteroids (except inhaled corticosteroids) during the previous month
* Treatment with diacerein, avocado and soya unsaponifiables, glucosamine sulphate or chondroitin sulphate, started in the previous 3 months, or irregular doses over the previous 3 months
* Hard of hearing (not being able to follow a telephone conversation properly)
* Patient without a telephone
* Pregnant women or nursing mothers
* Participation in other clinical studies, within 30 days before inclusion

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2012-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Patients assessment of WOMAC A1 pain when walking | 24 weeks

SECONDARY OUTCOMES:
Patients assessment of WOMAC A pain | 24 weeks
Patients assessment of WOMAC C function | 24 weeks
Patient global assessment | 24 weeks
OMERACT-OARSI responder rate | 24 weeks
Patient Acceptable Symptom State (PASS) | 24 weeks
Minimal Clinically Important Improvement (MCII) | 24 weeks
Adverse events observed or spontaneously reported by patients for each treatment | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Conrozier, MD, Principal Investigator — Lyon University Hospital (HCL)
Locations (17):
- France (16):
  - Cabinet Médical, Argeles
  - Centre Hospitalier de Belfort-Montbeliard, Belfort
  - Cabinet Médical, Billère
  - Cabinet Médical, Cabestany
  - Cabinet Médical Cabinet Médical, Cornebarrieu
  - Chu Henri Mondor, Créteil
  - Cabinet Médical, Lyon
  - Cabinet Médical, Metz
  - Hopital de Meulan-les-Mureaux, Meulan-en-Yvelines
  - Polyclinique Saint Odilon, Moulins
  - Centre Médical Europe, Paris
  - Institut de l'Appareil Locomoteur - Nollet, Paris
  - Hopitaux de Saint Marice, Saint-Maurice
  - Cabinet Médical, Strasbourg
  - Cabinet Medical, Valence
  - Cabinet Médical, Villeurbanne
- Hospital Princesse Grace de Monaco, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: Undecided